CLINICAL TRIAL: NCT02929160
Title: Optimal Method of Decompression of the Renal Collecting System in Acute Obstruction: a Prospective Randomised Trial
Brief Title: Percutaneous Nephrostomy Versus Stent In Sepsis Trial
Acronym: PERSIST
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: The Adelaide and Meath Hospital, incorporating The National Children's Hospital (Other)
Responsible Party: Principal Investigator, Rustom P Manecksha, MD, FRCS (Urol.), Consultant Urologist, The Adelaide and Meath Hospital, incorporating The National Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMNCH-GU-2016-1; 2016-004022-41 (EudraCT Number)
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Ureteric Calculus; Sepsis; Hydronephrosis
MeSH Terms: conditions — Ureterolithiasis; Sepsis; Hydronephrosis | interventions — Nephrostomy, Percutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCN (Experimental): Percutaneous nephrostomy
  Interventions: Procedure: Percutaneous nephrostomy
- JJ Stent (Experimental): Retrograde ureteric JJ stent
  Interventions: Procedure: Retrograde ureteric JJ stent

INTERVENTIONS:
Procedure: Percutaneous nephrostomy — Percutaneous nephrostomy tube insertion under radiological guidance
  Arms: PCN
Procedure: Retrograde ureteric JJ stent — Retrograde ureteric JJ stent insertion using cystoscopy
  Arms: JJ Stent

SUMMARY:
Randomized control trial to compare the efficacy and safety of percutaneous nephrostomy with retrograde ureteric stenting for emergency renal decompression in cases of obstruction and sepsis associated with ureteric calculi.

DETAILED DESCRIPTION:
The obstructed kidney in the setting of urosepsis is a urological emergency. Stone manipulation in the setting of active, untreated infection with concomitant urinary tract obstruction can lead to life-threatening sepsis. Therefore, urgent decompression of the collecting system is warranted.

There are two options for urgent decompression of an obstructed collecting system:

1. Image-guided percutaneous nephrostomy tube placement
2. Cystoscopic retrograde placement of a ureteric stent

This strategy allows drainage of infected urine and penetration of antibiotics to the affected renal unit. Definitive stone manipulation should be delayed until the infection is cleared following an appropriate course of antimicrobial therapy.

Both the European Association of Urology (EAU) and the American Urological Association (AUA) provide guidelines for management of an obstructed kidney. Both organisations provide evidence-based statements of the highest recommendation that urgent decompression of the kidney is mandated in the setting of sepsis. However, neither organisation recommend one decompression modality over the other. There is a lack of high quality up-to-date evidence to support a consensus view that one method of decompression is superior to the other.

This study aims to determine the most effective method of renal decompression in cases of obstruction and sepsis associated with ureteric calculi.

ELIGIBILITY:
Inclusion Criteria:

* Ureteric calculus with proximal hydronephrosis confirmed on CT KUB
* White cell count >12,000mm3 and/or temperature >38C

Exclusion Criteria:

* Uncorrected coagulopathy
* Urethral or ureteric stricture disease
* Urinary diversion
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Time to normalisation of white cell count and/or temperature | Within 1 week

SECONDARY OUTCOMES:
Length of hospital stay | Within 1 week

CONTACTS AND LOCATIONS:
Locations (2):
- Ireland (2):
  - The Adelaide and Meath Hospital, incorporating The National Children's Hospital, Tallaght, Dublin
  - St. James's Hospital, Dublin

IPD SHARING:
Plan to Share IPD: No